CLINICAL TRIAL: NCT02550574
Title: Use of 2-octylcyanoacrylate (Dermabond) During Cutaneous Wound Closure With Full-thickness Skin Grafts: a Randomized Split Wound Comparative Effectiveness Trial
Brief Title: Use of 2-octylcyanoacrylate With Full-thickness Skin Grafts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 773443
Record Dates: First submitted 2015-09-09; First posted 2015-09-15 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2016-12

CONDITIONS: Wound Closure Techniques
MeSH Terms: interventions — octyl 2-cyanoacrylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wound closure with 2-octylcyanoacrylate (Experimental): One side of the patient's wound defect will be assigned to wound closure with 2-octylcyanoacrylate liquid bonding agent).
  Interventions: Procedure: Wound Closure with 2-octylcyanoacrylate; Procedure: Wound Closure with 5-0 Vicryl Sutures
- Wound closure with 5-0 vicryl sutures (Active Comparator): One side of the patient's wound defect will be assigned to wound closure with 5-0 vicryl sutures.
  Interventions: Procedure: Wound Closure with 2-octylcyanoacrylate; Procedure: Wound Closure with 5-0 Vicryl Sutures

INTERVENTIONS:
Procedure: Wound Closure with 2-octylcyanoacrylate
Procedure: Wound Closure with 5-0 Vicryl Sutures

SUMMARY:
The purpose of this study is to determine whether the use of 2-octylcyanoacrylate during repair of cutaneous surgery wounds with full-thickness skin grafts improves scar cosmesis compared to wound closure with sutures.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether the use of 2-octylcyanoacrylate during repair of cutaneous surgery wounds with full-thickness skin grafts improves scar cosmesis compared to wound closure with sutures. Our aims are to compare outcomes using a split wound model, where half of the wound is treated with 2-octylcyanoacrylate and the other half is repaired with sutures, per the standard of care. Three-months post-surgery, the scar will be measured via the physician observer scar assessment scale, a validated scar instrument. Our hypothesis is that 2-octylcyanoacrylate will result in cosmetically superior wound outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Able to give informed consent themselves
* Patient scheduled for cutaneous surgical procedure with predicted closure with full-thickness skin graft
* Willing to return for follow-up visits

Exclusion Criteria:

* Mentally handicapped
* Unable to understand written and oral English
* Incarceration
* Under 18 years of age
* Pregnant Women
* Patients on systemic steroid therapies
* Patients with Marfans
* Patients with allergies to 2-octylcyanoacrylate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-12 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Appearance of Scar on the Patient and Observer Scar Assessment Scale | 3 months
  After surgical procedure, half of the subject's wound will be with 2-octylcyanoacrylate, while the other half is closed 5-0 vicryl sutures. After 3 months, subjects will return to clinic for evaluation of the cosmesis of both types of closure techniques.

SECONDARY OUTCOMES:
Incidence of Graft Failure on Case Report | 3 months
  The secondary endpoint will include incidence of graft failure (partial and complete on both sides).
Incidence of Complications on Case Report | 3 months
  Noting the presence or absence of bleeding, dehiscence, infection or spitting sutures.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Eisen, M.D., Principal Investigator — University of California, Davis